CLINICAL TRIAL: NCT01178827
Title: Sanctura Muscarinic Receptor Antagonist Resists Transport (SMART-II) Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA-SXR-09-005
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — trospium chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sanctura XR® (Experimental): Sanctura XR® (trospium chloride), 60mg once daily for 10 days
  Interventions: Drug: trospium chloride
- Oxybutynin IR (Active Comparator): Oxybutynin IR (oxybutynin immediate release), 5 mg three times daily for 2 days
  Interventions: Drug: oxybutynin IR
- Oxybutynin IR placebo (Placebo Comparator): Oxybutynin IR placebo three times daily for 2 days
  Interventions: Drug: oxybutynin IR placebo

INTERVENTIONS:
Drug: trospium chloride — trospium chloride (60mg) once daily for 10 days
  Other Names: Sanctura XR®
  Arms: Sanctura XR®
Drug: oxybutynin IR — oxybutynin IR (5 mg) three times daily for 2 days
  Arms: Oxybutynin IR
Drug: oxybutynin IR placebo — oxybutynin IR placebo three times daily for 2 days
  Arms: Oxybutynin IR placebo

SUMMARY:
This study will evaluate the cerebrospinal fluid levels of trospium chloride (Sanctura XR®) and oxybutynin immediate release (Oxybutynin IR) on memory performance in patients with overactive bladder and age associated memory impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents symptoms of overactive bladder
* Patient has age associated memory impairment
* No acute or unstable medical conditions

Exclusion Criteria:

* History of alcohol or substance abuse within 1 year prior to study
* Has donated in excess of 500mL of blood or plasma in the 30 days prior to study
* Has known bleeding disorder (hemophilia)
* Previous abdominal bypass surgery for obesity

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxybutynin IR: Oxybutynin IR (oxybutynin immediate release) 5 mg, three times daily for 2 days
Period: Overall Study
Arm/Group | Sanctura XR® | Oxybutynin IR | Oxybutynin IR Placebo
Started | 6 | 10 | 4
Completed | 6 | 10 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sanctura XR®: Sanctura XR® (60mg) once daily for 10 days
- Total: Total of all reporting groups
Arm/Group | Sanctura XR® | Oxybutynin IR | Oxybutynin IR Placebo | Total
Number analyzed (Participants) | 6 | 10 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.4 (6.3) | 68.3 (6.1) | 77.6 (12.3) | 72.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 2 | 11
  Male | 3 | 4 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Spinal Fluid Levels of Sanctura XR® at Day 10 Post-dose
Description: Cerebral spinal fluid levels of Sanctura XR® at Day 10 Post-dose. Cerebral spinal fluid is the fluid that surrounds the spinal cord and the inside of the brain. Samples were drawn from patients who received Sanctura XR®.
Time Frame: Day 10 Post-Dose
Population: All patients who received Sanctura XR®
Measure: Mean (Standard Deviation); unit: Nanograms (ng) per milliliter (mL)
Arm/Group | Sanctura XR® | Oxybutynin IR | Oxybutynin IR Placebo
Number analyzed (Participants) | 6 | 0 | 0
Nanograms (ng) per milliliter (mL) | NA (NA) — Below level of detection |  |

2. Primary Outcome: Cerebral Spinal Fluid Levels of Oxybutynin and N-Desethyl-Oxybutynin at Day 2 Post-dose
Description: Cerebral spinal fluid levels of Oxybutynin and N-Desethyl-Oxybutynin (metabolite of Oxybutynin) at Day 2 Post-dose. Cerebral spinal fluid is the fluid that surrounds the spinal cord and the inside of the brain. Samples were drawn from patients who received Oxybutynin IR.
Time Frame: Day 2 Post-Dose
Population: All patients who received Oxybutynin IR
Measure: Mean (Standard Deviation); unit: Nanograms (ng) per milliliter (mL)
Arm/Group | Sanctura XR® | Oxybutynin IR | Oxybutynin IR Placebo
Number analyzed (Participants) | 0 | 10 | 0
Nanograms (ng) per milliliter (mL)
  Oxybutynin |  | 0.0597 (0.0309) |
  N-Desethyl-Oxybutynin |  | 0.386 (0.235) |

3. Secondary Outcome: Plasma Levels of Sanctura XR® at Day 10 Post-dose
Description: Plasma levels of Sanctura XR® at Day 10 post-dose. Plasma is the liquid component of the blood in which the blood cells are suspended. Plasma samples were collected from each patient and analyzed for the drug the patient received.
Time Frame: Day 10 Post-Dose
Population: All patients who received of Sanctura XR®
Measure: Mean (Standard Deviation); unit: Nanograms (ng) per milliliter (mL)
Arm/Group | Sanctura XR® | Oxybutynin IR | Oxybutynin IR Placebo
Number analyzed (Participants) | 6 | 0 | 0
Nanograms (ng) per milliliter (mL) | 1.47 (1.03) |  |

4. Secondary Outcome: Plasma Levels of Oxybutynin and N-Desethyl-Oxybutynin at Day 2 Post-dose
Description: Plasma levels of Oxybutynin and N-Desethyl-Oxybutynin (metabolite of Oxybutynin) at Day 2 post-dose. Plasma is the liquid component of the blood in which the blood cells are suspended. Plasma samples were collected from each patient and analyzed for the drug the patient received.
Time Frame: Day 2 Post-Dose
Population: All patients who received of Oxybutynin IR
Measure: Mean (Standard Deviation); unit: Nanograms (ng) per milliliter (mL)
Arm/Group | Sanctura XR® | Oxybutynin IR | Oxybutynin IR Placebo
Number analyzed (Participants) | 0 | 10 | 0
Nanograms (ng) per milliliter (mL)
  Oxybutynin |  | 8.80 (2.84) |
  N-Desethyl-Oxybutynin |  | 47.0 (11.2) |

5. Secondary Outcome: Change From Baseline in Total Recall Score as Measured by the Hopkins Verbal Learning Test-Revised (HVLT-R) up to Day 10
Description: Change from Baseline in Total Recall Score as Measured by the HVLT-R up to Day 10. The HVLT-R is an instrument used to measure verbal learning and memory (recognition and recall). It consists of 3 learning trials: free recall, delayed recall, and yes/no delayed recognition. The total recall score was the sum of 3 'free recall' learning trials, and reflects the patient's ability to learn. The total score ranges from 0 (no memory) to 36 (best memory). A positive change from baseline indicates improved memory and a negative change from baseline indicates worsened memory.
Time Frame: Baseline, 10 Days
Population: Per Protocol: All subjects who completed the study.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Sanctura XR® | Oxybutynin IR | Oxybutynin IR Placebo
Number analyzed (Participants) | 6 | 10 | 4
Scores on a Scale
  Baseline | 22.5 (2.9) | 24.4 (3.3) | 24.0 (3.7)
  Change from Baseline up to Day 10 | -0.3 (3.3) | -3.3 (5.4) | -2.0 (4.8)

6. Secondary Outcome: Change From Baseline in Delayed Recall Score as Measured by the HVLT-R up to Day 10
Description: Change from Baseline in Delayed Recall Score as Measured by the HVLT-R up to Day 10. The HVLT-R is an instrument used to measure verbal learning and memory (recognition and recall). It consists of 3 learning trials: free recall, delayed recall, and yes/no delayed recognition. The total recall score was the sum of 3 'free recall' learning trials, and reflects the patient's ability to learn. The total score ranges from 0 (no memory) to 12 (best memory). A positive change from baseline indicates improved memory.
Time Frame: Baseline, 10 Days
Population: Per Protocol: All subjects who completed the study.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Sanctura XR® | Oxybutynin IR | Oxybutynin IR Placebo
Number analyzed (Participants) | 6 | 10 | 4
Scores on a Scale
  Baseline | 8.2 (1.2) | 9.4 (2.1) | 8.8 (2.1)
  Change from Baseline up to Day 10 | -1.2 (1.5) | -1.3 (1.6) | -0.3 (3.7)

7. Secondary Outcome: Change From Baseline in Total Recall Score as Measured by the Brief Visuospatial Memory Test-Revised (BVMT-R) up to Day 10
Description: Change from Baseline in total recall score as measured by the BVMT-R up to Day 10. The BVMT-R is an instrument used to measure visual learning and memory (recognition and recall). It consists of 3 learning trials: free recall, delayed recall, and yes/no delayed recognition trial. The total recall score is the sum of 3 free recall learning trials, and reflects the patient's ability to learn. The total score ranges from 0 (no memory) to 36 (best memory). A positive change from baseline indicates improved memory.
Time Frame: Baseline, 10 Days
Population: Per Protocol: All subjects who completed the study.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Sanctura XR® | Oxybutynin IR | Oxybutynin IR Placebo
Number analyzed (Participants) | 6 | 10 | 4
Scores on a Scale
  Baseline | 15.8 (6.6) | 20.3 (9.9) | 16.8 (11.3)
  Change from Baseline up to Day 10 | 1.2 (7.4) | -1.1 (5.3) | 0.0 (3.5)

8. Secondary Outcome: Change From Baseline in Delayed Recall Score as Measured by the BVMT-R up to Day 10
Description: Change from Baseline in delayed recall score as measured by the BVMT-R up to Day 10. The BVMT-R is an instrument used to measure visual learning and memory (recognition and recall). It consists of 3 learning trials: free recall, delayed recall, and yes/no delayed recognition trial. The total recall score is the sum of 3 free recall learning trials, and reflects the patient's ability to learn. The total score ranges from 0 (no memory) to 12 (best memory). A positive change from baseline indicates improved memory.
Time Frame: Baseline, 10 Days
Population: Per Protocol: All subjects who completed the study.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Sanctura XR® | Oxybutynin IR | Oxybutynin IR Placebo
Number analyzed (Participants) | 6 | 10 | 4
Scores on a Scale
  Baseline | 6.0 (4.2) | 8.0 (3.6) | 4.5 (5.3)
  Change from Baseline up to Day 10 | 0.2 (3.4) | -1.8 (3.5) | 2.3 (3.9)

ADVERSE EVENTS:
Arm/Group | Sanctura XR® | Oxybutynin IR | Oxybutynin IR Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10 | 0/4
Other Adverse Events (participants affected / at risk) | 5/6 | 7/10 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sanctura XR® (N=6) | Oxybutynin IR (N=10) | Oxybutynin IR Placebo (N=4)
Dry Mouth (Gastrointestinal disorders) | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 5 | 2
Lethargy (Nervous system disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Application Site Pruritus (General disorders) | 1 | 0 | 0
Body Temperature Increased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2
Dizziness (Nervous system disorders) | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Micturition Urgency (Renal and urinary disorders) | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.